CLINICAL TRIAL: NCT01136070
Title: A Prospective Study of Body Image, Social Avoidance and Distress and Psychological Functioning in Burn Patients
Status: Withdrawn | Type: Observational
Sponsor: Saint Elizabeth Regional Medical Center (Other)
Responsible Party: David Voigt, M.D., 555 South 70th Street Lincoln, NE 68510
Other Study IDs: 609-053
Record Dates: First submitted 2010-05-26; First posted 2010-06-03 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Depression; Anxiety; Body Image
Keywords: Psychological Functioning in Burn Patients
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Burn Trauma Patients

SUMMARY:
The present study seeks to examine the course of body image, social avoidance and psychosocial aspects of depression and anxiety over time in burn patients. Gaining a better understanding of the effects of burn injury on body image in burn patients over time could help us to better understand the psychosocial sequelae of burns and to identify potential interventions which may serve to improve the quality of life in burn patients.

DETAILED DESCRIPTION:
Gaining a better understanding of the effects of burn injury on body image in burn patients over time could help us to better understand the psychosocial sequelae of burns and to identify potential interventions which may serve to improve the quality of life in burn patients.

The original protocol has been modified to include more assessment times. The original protocol was set up to assess patients after patient discharge from the inpatient burn unit and at 6 and 12-months post discharge. The present protocol has been modified to capture assessments at 2 weeks, 3 months, 6 months, 9 months, 12 months post-burn. Patients will be assessed at these time points or until they are discharged from the outpatient burn clinic. In addition, inclusion criteria have been modified to include patients who are anticipated to have a follow-up visit to the burn outpatient clinic at 3 months post-burn. The original protocol required an anticipated follow-up for 12 months post-hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients are admitted to the Saint Elizabeth Regional Medical Center Burn Unit.
* Age 19 and older.
* Patients have the cognitive and physical capacity to answer the questionnaires.
* Patients are expected to be seen at follow-up clinic visits or if they are still in the hospital within 2 weeks and at 3 months (+ or - 4 weeks)post-burn.

Exclusion Criteria:

* Patients are unable to return for follow up visits

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Burn patients in community hospital with an estimated follow-up time of at least 3 months post-burn.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Satisfaction With Appearance Scale | 2 weeks post-burn
Brief Symptom Inventory | 2 weeks post-burn
Satisfaction with Appearance Scale | 3 months post-burn
Satisfaction with Appearance Scale | 6 months post-burn
  Data will be collected at this point only if subjects have not been discharged from the outpatient burn clinic.
Satisfaction with Appearance Scale | 9 months post-burn
  Data will be collected at this point only if subjects have not been discharged from the outpatient burn clinic.
Satisfaction with Appearance Scale | 12 months post-burn
  Data will be collected at this point only if subjects have not been discharged from the outpatient burn clinic.
Brief Symptom Inventory | 3 months post-burn
Brief Symptom Inventory | 6 months post-burn
  Data will be collected at this point only if subjects have not been discharged from the outpatient burn clinic.
Brief Symptom Inventory | 9 months post-burn
  Data will be collected at this point only if subjects have not been discharged from the outpatient burn clinic.
Brief Symptom Inventory | 12 months post-burn
  Data will be collected at this point only if subjects have not been discharged from the outpatient burn clinic.

SECONDARY OUTCOMES:
The Social Avoidance and Distress Scale | 2 weeks post-burn
The Social Avoidance and Distress Scale | 3 months post-burn
The Social Avoidance and Distress Scale | 6 moths post-burn
  Data will be collected at this point only if subjects have not been discharged from the outpatient burn clinic.
The Social Avoidance and Distress Scale | 9 months post-burn
  Data will be collected at this point only if subjects have not been discharged from the outpatient burn clinic.
The Social Avoidance and Distress Scale | 12 months post-burn
  Data will be collected at this point only if subjects have not been discharged from the outpatient burn clinic.

CONTACTS AND LOCATIONS:
Overall Officials: David W. Voigt, MD, Principal Investigator — Saint Elizabeth Regional Medical Center
Locations (1):
- Saint Elizabeth Regional Medical Center, Lincoln, Nebraska, United States